CLINICAL TRIAL: NCT04790123
Title: Adipose Tissue Injection for the Treatment of Complex Cryptoglandular Perianal Fistula
Acronym: AdiTiF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, Arantxa Muñoz-Duyos, Clinical Head of the General Surgery Service. Coloproctology Unit., Hospital Mutua de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P19/035
Record Dates: First submitted 2021-02-07; First posted 2021-03-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator)
  Interventions: Procedure: sham
- Experimental group (Experimental)
  Interventions: Procedure: Injection of autologous freshly collected adipose tissue

INTERVENTIONS:
Procedure: Injection of autologous freshly collected adipose tissue — injection of fresh autologous fat, previously lipoaspirates from the patient's abdomen and centrifugated, into the fistulous tract, after curettage and closure of the internal opening.
  Arms: Experimental group
Procedure: sham — curettage and closure of the internal orifice of the anal fistula and simulated intervention in the abdomen.
  Arms: Control group

SUMMARY:
The incidence of complex cryptoglandular anal fistula is high, it affects eminently young patients and implies an important alteration in their quality of life and high prevalence in sick leave. Its treatment remains a real challenge due to the limited efficacy of sphincter preservation techniques and the inevitable risk of faecal incontinence in those cases that require surgery. Goals: To evaluate the efficacy and safety of the injection of freshly collected autologous adipose tissue as a minimally invasive, highly reproducible alternative, without risk for the continence of the patient, and of very low cost, in the treatment of complex cryptoglandular anal fistula. Methodology: Prospective multicenter, randomized, double-blinded, parallel-group, placebo-controlled clinical trial. Randomization list for each center to ensure the balance of inter-center allocation. Patients older than 18 years with cryptoglandular anal fistula with suppuration for more than 6 weeks and less than 1 year, who have received at most: curettage and drainage placement will be included. Treatment group: injection of fresh autologous fat into the fistulous tract, after curettage and closure of the internal orifice, and after lipoaspirate fat in the abdomen and centrifugation thereof. Placebo group: curettage and closure of the internal orifice and simulated intervention in the abdomen. Evaluation: protocolized clinical history and fistula complexity score (CFS), subjective perception of its pathology, St.Marks continence score, Quality of life questionnaire (QoLAF), and endoanal 3D ultrasound, at baseline, at one week, and at 3, 6 and 12 months after the intervention. The patients and the evaluator will be blind to the treatment. Patients who cannot end up receiving treatment due to intraoperative incidents or medical decision will be excluded from the study (post randomization exclusion). In each center there will be a blind evaluator to perform the follow-ups and endoanal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Anal fistula with suppuration for more than 6 weeks and less than 1 year, that have not received any previous treatment or at most: curettage and drainage placement
* Complex cryptoglandular anal fistula: medium or high transsphincteric fistula, suprasphincteric fistula and extra sphincter fistula, shown by endoanal ultrasound.
* Low transsphincteric fistulas in patients with fecal incotinence.
* Any cryptoglandular anal fistula with risk factors for anal incontinence: anterior location fistula in women, history of pelvic surgery (hysterectomy, rectal resection), history of pelvic radiotherapy or previous anal surgery
* Draining with Seton placed >2 weeks before surgery and present at the time of treatment
* Disposition and ability to comply with the study protocol
* Signed informed consent

Exclusion Criteria:

* Patients diagnosed with inflammatory bowel disease
* Previous history of perianal fistula treated with any surgery different than curettage and seton placement (this include any type of surgery with curative intention, i.e. flap, lift technique, Radiofrequency, laser, stem cells, Filac, etc)
* Presence of Rectovaginal fistula
* Technical impossibility for lipoaspirate (liposuction) technique.
* Presence of perianal collections larger than 2cm
* Presence of several paths from 1 internal hole only
* Presence of secondary fistula paths or tracts
* Perianal surgery necessary at the time of planning the fistula treatment, for reasons other than fistula.
* Major surgery needed within 28 days of recruitment
* Immunomodulator treatment or corticotherapy in a previous period of 6 months
* Stoma patients
* Serious medical or psychiatric illness that requires frequent hospitalization.
* Pregnancy, pregnancy plans or breastfeeding in the next 12 months
* Active smokers, or ex-smokers of less than 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-11-14 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Complete fistula healing | 24 weeks
  Comparison of the proportion of cases with complete fistula healing within 24 weeks of the intervention, defined as the absence of drainage through the external orifice, its complete reepithelialization and the absence of collections confirmed by endoanal ultrasound.

SECONDARY OUTCOMES:
Patient's Quality of life | 6 and 12 months after treatment.
  Improvement in quality of life (measured with the Quality of Life in Patients with Anal Fistula Questionnaire, QoLAF).
  Score from 14 to 70, where 14 means "no quality of life alteration" and 70 means "severe quality of life alteration".
Patient's Subjective Perception | 6 and 12 months after treatment.
  Improvement in patient subjective evaluation using a Visual Analogue Scale (VAS).
  Score from 0 to 10, where 0 means "no problem" and 10 means "severe problem and alteration of my quality of life".
Fistula severity | 6 and 12 months after treatment.
  Improvement in fistula severity according to the Complexity Fistula score (CFS).
  Score from 3 to 15, where 3 means "low complexity" and 15 means "high complexity"
Adverse events | 3, 6 and 12 months after treatment.
  Evaluation of the safety by the incidence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No